CLINICAL TRIAL: NCT00379106
Title: Arm Function and Quality of Life Following Mastectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Kathy Dieruf, MD; Principal Investigator, Universtiy of New Mexico - CRTC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1002C
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer
Keywords: Supportive; Mastectomy; Quality of Life; Arm Function
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group1 (Active Comparator)
  Interventions: Procedure: Arm exercises.
- Group 2 (Experimental)
  Interventions: Procedure: Arm Exercises

INTERVENTIONS:
Procedure: Arm exercises. — Basic active exercise program at home.
  Arms: Group1
Procedure: Arm Exercises — Instruction in the same active exercise program along with additional exercises using exercise equipment and stretching exercises
  Arms: Group 2

SUMMARY:
To measure arm function and quality of life of mastectomy patients.

DETAILED DESCRIPTION:
Treatment: Randomized to one of two treatment arms. Group One: Basic active exercise program at home. Group Two: Instruction in the same active exercise program along with additional exercises using exercise equipment and stretching exercises. Range of Motion measurements will be taken at the first session, 1 month, 6 weeks, 3 months, 6 months and 1 year. Patients will complete demographic form, functional questionnaire, and QOL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been referred from UNMH to CRTC for further treatment following mastectomy/lumpectomy surgery.

Exclusion Criteria:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-10; Primary Completion 2005-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Arm Function and Quality of Life Following Mastectomy | Motion measurements will be taken at the first session, 1 month, 6 weeks, 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Dieruf, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States